CLINICAL TRIAL: NCT01658839
Title: An Open-Label, Pharmacokinetic and Safety Study of Travoprost Ophthalmic Solution, 0.004% in Pediatric Glaucoma or Ocular Hypertension Patients
Brief Title: Pharmacokinetic and Safety Study of Travoprost 0.004% in Pediatric Glaucoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-12-009; 2012-001640-22 (EudraCT Number)
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: pediatric glaucoma; pediatric ocular hypertension; travoprost
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Hydrophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Travoprost (Experimental): Travoprost ophthalmic solution, 0.004% (new formulation), one drop administered topically in the inferior cul-de-sac of the eye each morning at 9 AM (± 60 minutes) for 7 days
  Interventions: Drug: Travoprost ophthalmic solution, 0.004% (new formulation)

INTERVENTIONS:
Drug: Travoprost ophthalmic solution, 0.004% (new formulation) — Travoprost ophthalmic solution, 0.004%, new formulation

SUMMARY:
The purpose of this study was to assess the safety and describe the steady-state plasma pharmacokinetic (PK) profiles of Travoprost ophthalmic solution, 0.004% (new formulation) following a once daily administration for 7 days in pediatric glaucoma or ocular hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma or ocular hypertension in at least 1 eye.
* Parent/legal guardian must provide informed consent, and children must agree to sign an approved assent form when applicable.
* Must agree to comply with the requirements of the study and must be accompanied by a parent/guardian.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential that are currently pregnant, have a positive result on a pregnancy test at the Screening Visit, intend to become pregnant during the study period, are breast feeding, or are not using birth control measures.
* One sighted eye or monocular, including patients who cannot be dosed in both eyes for any reason.
* History of chronic, recurrent or severe inflammatory eye disease.
* Ocular trauma requiring medical attention within the past 3 months prior to the Screening Visit.
* Ocular infection or ocular inflammation within the past 30 days prior to the Screening Visit.
* Clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment.
* Other severe ocular pathology (including severe dry eye), that in the opinion of the Investigator, would preclude the administration of a topical prostaglandin analogue.
* Intraocular surgery within the past 30 days prior to the Screening Visit.
* Any abnormality preventing reliable tonometry.
* Any other conditions including severe illness which would make the patient, in the opinion of the Investigator, unsuitable for the study.
* Hypersensitivity to prostaglandin analogues or to any component of the study medications in the opinion of the Investigator.
* Therapy with another investigational agent or device within 30 days prior to the Screening Visit.
* Body weight < 5kg.
* Other protocol-defined exclusion criteria may apply.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subha Venkataraman, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 investigational centers located in the US, 1 located in France, 1 located in Spain, and 1 located in Saudi Arabia.
Pre-assignment Details: Twenty-five participants were enrolled and completed the study. This reporting group includes all enrolled participants (25).
Period: Overall Study
Arm/Group | Travoprost
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled participants.
Arm/Group | Travoprost
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Travoprost Free Acid Plasma Concentration (Cmax)
Description: Travoprost free acid plasma concentrations at each collection time point (predose, 10, 20, 40, 80 minutes postdose) were quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS). Cmax was calculated for each participant with at least 1 quantifiable time point.
Time Frame: Day 7, Up to 80 minutes postdose
Population: This analysis group includes all participants who received at least 2 doses of the study drug, satisfied protocol required criteria relevant to the assessments of PK parameters, had at least 1 postdose blood draw, and for whom adequate PK data were collected (without collection or analytical deviations that would affect the integrity of the data).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Travoprost
Number analyzed (Participants) | 11
ng/mL
  Overall (n=11) | 0.0256 (0.0158)
  2 mo to < 3 years (n=2) | 0.0471 (0.0105)
  3 to <12 years (n=6) | 0.0258 (0.0128)
  12 to <18 years (n=3) | 0.0109 (0.000046)

2. Primary Outcome: Time to Reach Cmax (Tmax)
Description: Analyte plasma concentrations at each collection time point (predose, 10, 20, 40, 80 minutes postdose) were quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS). Tmax was calculated for each participant with at least 1 quantifiable time point.
Time Frame: Day 7, Up to 80 minutes postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Travoprost
Number analyzed (Participants) | 11
hours
  Overall (n=11) | 0.25 (0.15)
  2 mo to <3 years (n=2) | 0.26 (0.11)
  3 to <12 years (n=6) | 0.17 (0.00)
  12 to <18 years (n=3) | 0.39 (0.26)

3. Primary Outcome: Time to Last Measurable Concentration (Tlast)
Description: Analyte plasma concentrations at each collection time point (predose, 10, 20, 40, 80 minutes postdose) were quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS). Tlast was calculated for each participant with at least 1 quantifiable time point.
Time Frame: Day 7, Up to 80 minutes postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Travoprost
Number analyzed (Participants) | 11
hours
  Overall (n=11) | 0.42 (0.35)
  2 mo to <3 years (n=2) | 0.34 (0.01)
  3 to <12 years (n=6) | 0.46 (0.47)
  12 to <18 years (n=3) | 0.39 (0.26)

4. Primary Outcome: Area Under the Analyte Plasma Concentration-time Curve to the Last Quantifiable Sampling Time Point [AUC(0-tlast)]
Description: Analyte plasma concentrations at each collection time point (predose, 10, 20, 40, 80 minutes postdose) were quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS). AUC(0-tlast) was calculated for each participant with at least 2 quantifiable time points.
Time Frame: Day 7, Up to 80 minutes postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Travoprost
Number analyzed (Participants) | 6
ng*hr/mL
  Overall (n=6) | 0.0116 (0.0099)
  2 mo to <3 years (n=2) | 0.0101 (0.0014)
  3 to <12 years (n=4) | 0.0123 (0.0127)

5. Primary Outcome: Area Under the Analyte Plasma Concentration-time Curve Over the Dosing Interval (Inf)[AUC(0-∞)]
Description: Analyte plasma concentrations at each collection time point (predose, 10, 20, 40, 80 minutes postdose) were quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS). AUC(0-∞) was calculated for each participant with at least 3 quantifiable time points.
Time Frame: Day 7, Up to 80 minutes postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Travoprost
Number analyzed (Participants) | 1
ng*hr/mL
  Overall (n=1) | 0.0389 (NA) — Standard deviation was not estimated
  3 to <12 years (n=1) | 0.0389 (NA) — Standard deviation was not estimated

6. Primary Outcome: Half-life (t½)
Description: Analyte plasma concentrations at each collection time point (predose, 10, 20, 40, 80 minutes postdose) were quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS). T½ was calculated for each participant with at least 3 quantifiable time points.
Time Frame: Day 7, Up to 80 minutes postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Travoprost
Number analyzed (Participants) | 1
hours
  Overall (n=1) | 0.53 (NA) — Standard deviation was not estimated
  3 to <12 years (n=1) | 0.53 (NA) — Standard deviation was not estimated

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (6 months). This analysis group includes all participants who received study drug.
Description: An AE is defined as any untoward medical occurrence in a participant who is administered a study medication, regardless of whether or not the event has a causal relationship with the medication. Reports of AEs were obtained as solicited comments from the study participants and as observations by the study Investigator.
Arm/Group | Travoprost
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Travoprost (N=25)
Trabeculectomy (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.